CLINICAL TRIAL: NCT06128460
Title: Adjuvant Chemoradiotherapy Followed by Zimberelimab for Locally Advanced Cervical Cancer (IB3, IIA2) Patients
Brief Title: Adjuvant Chemoradiotherapy Followed by Zimberelimab for Locally Advanced Cervical Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Keqin Hua, Director of Gynecological Oncology, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLS-010-672
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — zimberelimab; Platinum; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concurrent themoradiotherapy Followed by Zimberelimab (Experimental): 1. Radiotherapy: Intensity modulated conformal radiation therapy (IMRT) is used for external irradiation, and the pelvic target volume dose (PTV) is: 45-50 Gy/1.8Gy/25-28f; the stump margin is positive, and after the external irradiation is completed, Additional CT-guided three-dimensional conformal brachytherapy, HR-CTV: 24--30Gy/4-5f.
  2. Concurrent chemotherapy: performed during external radiotherapy. Starting from the first week of radiochemotherapy, cisplatin 40 mg/m2 was given. Chemotherapy is given every 7 days, up to 5-6 times;
  3. Zimberelimab injection: 240 mg/time, intravenous infusion, administered every 21 days, starting within four weeks after completing concurrent chemoradiotherapy, and maintained for 8 cycles
  Interventions: Drug: Zimberelimab; Drug: Platinum; Radiation: radiotherapy

INTERVENTIONS:
Drug: Zimberelimab — 240mg, q3w，8 cycles
Drug: Platinum — cisplatin 40mg/m2 for 5-6 cycles
Radiation: radiotherapy — 45-50Gy/1.8Gy/25-28f

SUMMARY:
Locally advanced cervical cancer (stage IB3, IIA2) patients with postoperative risk factors need better treatment. We initiated a clinical study to explore the effectiveness of adjuvant chemoradiotherapy followed by Zimberelimab for these patients.

DETAILED DESCRIPTION:
For cervical cancer, although clinical research on PD-1 monoclonal antibodies was launched relatively late, the research results so far show that PD-1 monoclonal antibodies combined with chemotherapy have a high clinical effectiveness and a relatively high efficacy in the treatment of advanced/recurrent cervical cancer. Good security. However, there is currently a lack of clinical evidence for the use of PD-1 monoclonal antibodies combined with chemoradiotherapy in the treatment of high-risk patients after cervical cancer surgery. Therefore, this study intends to explore the clinical efficacy of postoperative adjuvant radiochemotherapy followed by PD-1 monoclonal antibody in the treatment of high-risk patients with locally advanced (IB3, IIA2) cervical cancer after surgery, and provide a new solution for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervical squamous cell carcinoma, cervical adenocarcinoma, or cervical adenosquamous carcinoma;
* According to FIGO2018 staging, patients with locally advanced cervical cancer (IB3, IIA2) who require concurrent radiotherapy and chemotherapy;
* Patients with radical surgery for cervical cancer;
* Female patients: 18-70 years old;
* ECOG physical condition score: 0~1 point;
* Subjects have not received previous immunotherapy;
* Expected survival ≥6 months;
* Women of reproductive age should agree to use contraceptives (such as Iuds, contraceptives, or condoms) during the study period and for 6 months after the study ends; Have a negative serum or urine pregnancy test within 7 days prior to study enrollment and must be a non-lactating patient;
* For adequate organ function as defined in the protocol, test samples must be collected within 7 days prior to initiation of the study therapy
* Subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Subjects have histological subtypes other than those permitted by inclusion criteria;
* Severe hypersensitivity to cepalizumab and/or any of its excipients (≥ grade 3);
* Participate in or have participated in other clinical trials within 4 weeks before enrollment;
* Have received or will receive inactivated vaccine within 30 days prior to the first study treatment;
* Received a combination of systemic immune stimulants, colony-stimulating factors, interferon, interleukin, and vaccine within 6 weeks or 5 half-lives (if shorter) prior to initial administration;
* Have been diagnosed with an immune deficiency or are receiving chronic systemic steroid therapy (doses greater than 10mg daily equivalent of prednisone) or any other form of immunosuppressive therapy within 7 days prior to the first dose;
* Have an active autoimmune disease in the past 2 years that requires systemic treatment (such as the use of disease-modulating drugs, corticosteroids, or immunosuppressive drugs);
* Have a history of (non-infectious) pneumonia requiring steroid treatment or have a current (non-infectious) pneumonia;
* An active infection requiring systematic treatment;
* Known history of HIV infection;
* A known history of hepatitis B (defined as HBsAg reactive) or known active hepatitis C virus (defined as detection of HCV RNA[qualitative]) infection;
* Known active tuberculosis (TB; Tuberculosis) medical history;
* Has received allogeneic tissue/solid organ transplantation;
* Suffering from central nervous system metastases such as brain metastases;
* Patients with uncontrolled chest and abdominal fluid;
* Patients with mobility disorders such as pathological fractures caused by tumor bone metastasis;
* Insufficient hematopoietic function of bone marrow;
* Abnormal liver;
* Abnormal kidney;
* Bleeding risk;
* Cardiovascular and cerebrovascular abnormalities.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
changes in tumor-related biomarkers | 3 years
  changes of tumor- related biomarkers (T cell receptor library profile and peripheral blood ctDNA content analysis)

SECONDARY OUTCOMES:
OS | 5 years
  Overall Survival
DFS | 2 years
  Disease Free Survival
AE | 3 years
  Adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Keqin Hua, Doctor, Principal Investigator — Gynecology and obstetrics hospital of fudan university

IPD SHARING:
Plan to Share IPD: No